CLINICAL TRIAL: NCT02614885
Title: Feasibility Study of Cavitary Radiofrequency Ablation in Excised Mastectomy Breast Tissue
Status: Completed | Type: Observational
Sponsor: Innoblative Designs, Inc. (Industry)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-01
Record Dates: First submitted 2015-11-20; First posted 2015-11-25 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Prophylactic Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prophylactic Mastectomy: Females undergoing prophylactic mastectomy with RFA performed on the excised tissue.
  Interventions: Device: RFA

INTERVENTIONS:
Device: RFA — Radiofrequency ablation of the cavity walls of a simulated lumpectomy in the excised prophylactic mastectomy tissue.

SUMMARY:
This is a single-arm, prospective study of a radiofrequency ablation device on the excised breast tissue of ten (10) prophylactic mastectomy patients. The ablation lesion created by the device will be analyzed histologically.

DETAILED DESCRIPTION:
This study is a single-center, prospective, open label study of a radiofrequency ablation device. 10 patients who are scheduled to undergo prophylactic mastectomy will be recruited by the clinical investigators at the investigational site in accordance with the inclusion and exclusion criteria. Once the breast tissue is removed, the radiofrequency ablation device will be used on the ex vivo tissue to ablate a lesion around a cavity created in the tissue. The ablation lesion will be characterized. The study period per subject is the time it takes to assess the ablation lesion histologically.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. At least 18 years of age
3. Scheduled to receive a standard of care prophylactic mastectomy (or prophylactic bi-lateral mastectomy)
4. The patients' breast(s) to be included in the study are undiseased
5. The patient has adequate breast volume for ex vivo ablation procedure

Exclusion Criteria:

1. The patient is receiving a skin sparing mastectomy(s)
2. The patient has had previous exposure to chemotherapy or radiation therapy
3. The patient has implants in the breast(s) to be included in the study
4. The patient is currently pregnant or lactating
5. The patient has tissue markers implanted in the breast to be included in the study (unless these can be removed when creating a cavity in the ex vivo breast tissue)
6. The patient has had previous surgery on the breast(s) to be included in the study (unless study investigator determines that this will not affect the validity of data in this study)
7. The patient in participating in any other clinical study of a device or drug that may impact the participant safety of the validity of data acquired in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for prophylactic mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Histologic measurement of cavitary ablation lesions created by the Innoblative radiofrequency ablation device in ex vivo breast tissue to correlate ablation size with ablation parameters. | Two weeks after surgery
  Histologic analysis of ablation depth around the cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela A Ochoa, MD, Principal Investigator — UAMS